CLINICAL TRIAL: NCT04159077
Title: Reduction of Post-Operative Urinary Retention With Tamsulosin Versus Placebo (REPOURT- P) Trial
Acronym: REPOURT-P
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SJHH_REPOURT_P
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-01

CONDITIONS: Urinary Catheterization; Thoracic Surgery; Thoracic Epidural Analgesia
Keywords: Post-operative urinary retention; Tamsulosin; urinary tract infections; catheter
MeSH Terms: conditions — Urinary Tract Infections | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamsulosin Hydrochloride (HCL) (Experimental): Consenting patients undergoing pulmonary resection will receive a 5-day allotment of tamsulosin HCL to be started 3 days prior to their date of surgery.
  Interventions: Drug: Tamsulosin Hydrochloride
- Placebo (Placebo Comparator): Consenting patients undergoing pulmonary resection will receive a 5-day allotment of placebo to be started 3 days prior to their date of surgery.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tamsulosin Hydrochloride — Tamsulosin HCL is an alpha blocker. It relaxes the muscles in the prostate and bladder neck, making easier to urinate. The dosage used will be 0.4 mg (administered once daily)
  Other names: Flomax
  Arms: Tamsulosin Hydrochloride (HCL)
Drug: Placebos — Half of the patients will be assigned to receive placebo tablets in the same manner as the active intervention. These tablets will have no effect.
  Arms: Placebo

SUMMARY:
The purpose of this study are to determine the efficacy of tamsulosin compared to placebo in reducing post-operative urinary retention and improving other clinical outcomes in people undergoing thoracic surgery.

DETAILED DESCRIPTION:
Post-operative urinary retention (POUR) is not an uncommon complication following thoracic surgery. It has been reported to occur in up to 12-67% of patients with the use of thoracic epidural analgesia1. Risk factors associated with urinary retention in thoracic patients include male, age over 40 years, type 2 diabetes, undergoing lung resection and the use of thoracic epidural analgesia2. Patients who experience urinary retention are treated with a straight catheter and may subsequently require the placement of an indwelling catheter. The use of these catheters is associated with numerous complications. The best studied complications are infectious and include catheter associated urinary tract infections (CAUTIs). However, many patients continue to experience symptoms well after their catheters have been removed.

Tamsulosin is an alpha one adrenergic receptor blocked that is indicated for the treatment of lower urinary tract symptoms in the context of benign prostatic hyperplasia. However, it is often used in clinical practice to treat other pathologies such as acute urinary retention and nephrolithiasis.

The objectives of this study are to determine the efficacy of tamsulosin compared to placebo in reducing post-operative urinary retention and catheter related complications in people undergoing thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients greater than the age of 40 and/or with type 2 diabetes undergoing pulmonary surgery who did not undergo straight or indwelling urinary catheterization intraoperatively.

   OR
2. Male patients receiving a thoracic epidural analgesia undergoing pulmonary surgery who did not undergo straight or indwelling urinary catheterization intraoperatively

Exclusion Criteria:

1. Active treatment of Benign Prostatic Hyperplasia (BPH)
2. Hypersensitivity or allergy to tamsulosin HCL
3. Active treatment with tamsulosin or other alpha-blocker or uses of tamsulosin/ other alpha-blocker within 3 weeks of enrollment date
4. Active urinary tract infection
5. History of urological disorder specified as urethral stricture, BPH, bladder or prostate malignancy
6. History of urological surgery (Transurethral resection of the Prostate, Transurethral resection of the Bladder, Bladder suspension, prostatectomy)
7. Underlying neurological disorders resulting in impaired bladder function
8. Any known contraindication to the use of tamsulosin HCL

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 350 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of post-operative urinary retention (POUR) | 0-24 hours
  Rate of POUR; defined as requiring straight or indwelling catheterization at any point in the post-operative period.

SECONDARY OUTCOMES:
Rate and number of straight catheterizations | 0-7 days
  Rate and number of straight catheterizations
Rate of indwelling catheterization | 0-7 days
  Rate of indwelling catheterization
Time to first catheterization | 0-24 hours
  Time to first catheterization
Treatment emergent Adverse Events | -3 days to 2 days
  Treatment emergent Adverse Events as reported by the FDA (the Federal Drug Administration )
Rates of catheter complications within 30 days of catheterization | 0 to 30 days
  e.g. CAUTI, Urethral Trauma, Hematuria, urethral stricture
Duration of hospital length of stay | 0 to 365 days
  Date of admission to date of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Shargall, MD, PhD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeung JH, Gates S, Naidu BV, Wilson MJ, Gao Smith F. Paravertebral block versus thoracic epidural for patients undergoing thoracotomy. Cochrane Database Syst Rev. 2016 Feb 21;2(2):CD009121. doi: 10.1002/14651858.CD009121.pub2. PMID 26897642
- [Background] Kim KW, Lee JI, Kim JS, Lee YJ, Choi WJ, Jung H, Park KY, Park CH, Son KH. Risk factors for urinary retention following minor thoracic surgery. Interact Cardiovasc Thorac Surg. 2015 Apr;20(4):486-92. doi: 10.1093/icvts/ivu445. Epub 2015 Jan 6. PMID 25564576
- [Background] Saint S, Trautner BW, Fowler KE, Colozzi J, Ratz D, Lescinskas E, Hollingsworth JM, Krein SL. A Multicenter Study of Patient-Reported Infectious and Noninfectious Complications Associated With Indwelling Urethral Catheters. JAMA Intern Med. 2018 Aug 1;178(8):1078-1085. doi: 10.1001/jamainternmed.2018.2417. PMID 29971436
- [Background] Shokrpour M, Shakiba E, Sirous A, Kamali A. Evaluation the efficacy of prophylactic tamsulosin in preventing acute urinary retention and other obstructive urinary symptoms following colporrhaphy surgery. J Family Med Prim Care. 2019 Feb;8(2):722-727. doi: 10.4103/jfmpc.jfmpc_18_19. PMID 30984702
- [Background] Basheer A, Alsaidi M, Schultz L, Chedid M, Abdulhak M, Seyfried D. Preventive effect of tamsulosin on postoperative urinary retention in neurosurgical patients. Surg Neurol Int. 2017 May 10;8:75. doi: 10.4103/sni.sni_5_17. eCollection 2017. PMID 28584678